CLINICAL TRIAL: NCT01925417
Title: A Phase 2 Open-label Clinical Trial Demonstrating the Safety of RBX2660 Microbiota Suspension for the Treatment of Recurrent Clostridium Difficile-associated Diarrhea (CDAD): the PUNCH CD Study
Brief Title: Microbiota Restoration Therapy for Recurrent Clostridium Difficile-associated Diarrhea
Acronym: PUNCH CD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rebiotix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-001
Record Dates: First submitted 2013-08-15; First posted 2013-08-19 (Estimated); Results first posted 2015-07-01 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2018-09

CONDITIONS: Recurrent Clostridium Difficile Infection
Keywords: Clostridium difficile; C diff; Microbiota Restoration Therapy; MRT; microbiota suspension; CDI; CDAD; Fecal transplant; Fecal Microbiota Transplant; FMT; Diarrhea; Fecal bacteriotherapy
MeSH Terms: conditions — Clostridium Infections; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RBX2660 (microbiota suspension) (Experimental): enema-based delivery of RBX2660
  Interventions: Biological: RBX2660 (microbiota suspension)

INTERVENTIONS:
Biological: RBX2660 (microbiota suspension)

SUMMARY:
This study will assess the safety of a new biologic drug, RBX2660 (microbiota suspension) as a treatment for recurrent Clostridium difficile-associated diarrhea (CDAD), which is the primary symptom of recurrent Clostridium difficile infection. All eligible subjects will receive RBX2660.

DETAILED DESCRIPTION:
This is the first study of a microbiota suspension derived from intestinal microbes. The primary assessments for this open label, multi-center study are (i) occurrence of product-related adverse events and (ii) resolution of CDAD at 56 days after administration of RBX2660. Subjects will also be assessed for time to CDAD recurrence, quality of life changes, and number of hospitalizations and length of stay for recurrent CDAD. Study visits will be at 7, 30, and 60 days after RBX2660 administration with additional follow-up at 3 and 6 months post treatment. Patients who have had at least two recurrences of CDAD after a primary episode and have completed at least two rounds of standard-of-care oral antibiotic therapy or have had at least two episodes of severe CDAD resulting in hospitalization may be eligible for the study.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Medical record documentation of CDAD either: a) at least two recurrences after a primary episode and have completed at least two rounds of standard-of-care oral antibiotic therapy or b) have had at least two episodes of severe CDAD resulting in hospitalization.
* Willing and able to have an enema(s).
* Already taking or will start a course of oral antibiotics for CDAD symptoms for 10-14 days, including at least seven days of oral vancomycin.
* Willing and able to complete the required subject diary.

Exclusion Criteria:

* Continued (uncontrolled) CDAD after completing a 10-14 day course of oral antibiotics.
* Requires antibiotic therapy for a condition other than CDAD.
* Previous fecal transplant prior to study enrollment.
* History of inflammatory bowel disease (IBD), e.g., ulcerative colitis, Crohn's disease, or microscopic colitis.
* History of irritable bowel syndrome (IBS).
* History of chronic diarrhea.
* History of celiac disease.
* History of cirrhosis of the liver or ascites.
* Disease symptoms caused by a confirmed intestinal pathogen other than Clostridium difficile.
* Has a colostomy.
* Intraabdominal surgery within the last 60 days.
* Evidence of active, severe colitis.
* History of short gut syndrome or motility disorders.
* Requires the regular use of medications that affect bowel motility (e.g., metoclopramide, narcotics, loperamide).
* Planned therapy in the next 3 months that may cause diarrhea (e.g., chemotherapy).
* Planned surgery requiring perioperative antibiotics within 6 months of study enrollment.
* Life expectancy of < 12 months.
* Compromised immune system, e.g., HIV infection (any CD4 count); AIDS-defining diagnosis or CD4 <200/mm3; inherited/primary immune disorders; immunodeficient or immunosuppressed due to a medical condition or medication; current or recent (< 90 days) treatment with chemotherapy; or current or recent (< 90 days) treatment with immunosuppressant medications.
* Taking steroids (≥ 20 mg a day) or is expected to be on steroids for more than 30 days after enrollment.
* Neutropenia (white blood cell count <1000 cells/µL).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Drekonja, MD, Study Chair — Veteran Administration Medical Center
Locations (13):
- United States (13):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Denver Health and University of Colorado, Denver, Colorado
  - Borland-Groover Clinic, Jacksonville, Florida
  - Edward Hines Jr VA Hospital (veterans only), Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Ochsner Clinic, New Orleans, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Detroit Medical Center, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Sanford Research/USD, Fargo, North Dakota

REFERENCES:
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Gough E, Shaikh H, Manges AR. Systematic review of intestinal microbiota transplantation (fecal bacteriotherapy) for recurrent Clostridium difficile infection. Clin Infect Dis. 2011 Nov;53(10):994-1002. doi: 10.1093/cid/cir632. PMID 22002980
- [Background] Rohlke F, Stollman N. Fecal microbiota transplantation in relapsing Clostridium difficile infection. Therap Adv Gastroenterol. 2012 Nov;5(6):403-20. doi: 10.1177/1756283X12453637. PMID 23152734
- [Derived] Lee C, Feuerstadt P, Louie T, Bancke L, Guthmueller B, Harvey A, Hoeyer F, Orenstein R, Dubberke ER, Khanna S. Integrated analysis of the safety of fecal microbiota, live-jslm in adults with recurrent Clostridioides difficile infection from five prospective clinical trials: an update. Therap Adv Gastroenterol. 2025 Nov 12;18:17562848251395566. doi: 10.1177/17562848251395566. eCollection 2025. PMID 41245385
- [Derived] Langdon A, Schwartz DJ, Bulow C, Sun X, Hink T, Reske KA, Jones C, Burnham CD, Dubberke ER, Dantas G; CDC Prevention Epicenter Program. Microbiota restoration reduces antibiotic-resistant bacteria gut colonization in patients with recurrent Clostridioides difficile infection from the open-label PUNCH CD study. Genome Med. 2021 Feb 16;13(1):28. doi: 10.1186/s13073-021-00843-9. PMID 33593430
- [Derived] Orenstein R, Dubberke E, Hardi R, Ray A, Mullane K, Pardi DS, Ramesh MS; PUNCH CD Investigators. Safety and Durability of RBX2660 (Microbiota Suspension) for Recurrent Clostridium difficile Infection: Results of the PUNCH CD Study. Clin Infect Dis. 2016 Mar 1;62(5):596-602. doi: 10.1093/cid/civ938. Epub 2015 Nov 12. PMID 26565008

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from 07/15/13 to 12/16/13 at 13 medical clinics in the United States. Recruiment was performed by trained investigators and study coordinators.
Groups:
- RBX2660 (Microbiota Suspension): This was an open-label, non-randomized, non-controlled subjects. All treated subjects received RBX2660 (microbiota suspension).
Period: Overall Study
Arm/Group | RBX2660 (Microbiota Suspension)
Started | 34
Completed | 31
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- RBX2660 (Microbiota Suspension): Open-label; all subjects received RBX2660
Arm/Group | RBX2660 (Microbiota Suspension)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 66.8 [26.7 to 89.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Serious Adverse Events Through 56 Days After the Last Treatment With RBX2660
Description: Safety will be assessed by evaluating the incidence of serious adverse events through 56 days after the last treatment with RBX2660.
Time Frame: 56 days
Population: 31 subjects had evaluable data at 56 days.
Measure: Number; unit: number of reported SAEs through 56 days
Arm/Group | RBX2660 (Microbiota Suspension)
Number analyzed (Participants) | 31
number of reported SAEs through 56 days | 10

2. Secondary Outcome: Long-term Safety
Description: The incidence of serious adverse events will be assessed through 6 months after the last treatment with RBX2660.
Time Frame: 6 months
Population: 31 subjects had evaluable data at 6 months.
Measure: Number; unit: number of reported SAEs
Arm/Group | RBX2660 (Microbiota Suspension)
Number analyzed (Participants) | 31
number of reported SAEs | 20

3. Secondary Outcome: Absence of CDAD at 56 Days
Description: Number of participants who were determined to be free of CDAD at Day 56 after receiving their last dose of RBX2660.
Time Frame: 56 days
Population: 31 subjects had evaluable data at 56 days.
Measure: Number; unit: participants with treatment success
Arm/Group | RBX2660 (Microbiota Suspension)
Number analyzed (Participants) | 31
participants with treatment success | 27

4. Secondary Outcome: Quality of Life (SF-36)
Description: Quality of Life (SF-36) will be assessed by comparing the subject's baseline quality of life score to his/her scores obtained at the 7-, 30- and 60-day follow-up visits.
  The scale is from 0-100, with higher scores meaning better outcomes.
Time Frame: 60 days
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- RBX2660 (Microbiota Suspension): RBX2660 (microbiota suspension) enema-based delivery
Arm/Group | RBX2660 (Microbiota Suspension)
Number analyzed (Participants) | 34
score on a scale
  Baseline | 42.2 (14.6)
  7-Day | 47.7 (11.7)
  30-DAy | 48.6 (11.8)
  60-Day | 51.3 (11.2)

5. Secondary Outcome: Post-treatment Hospitalization Data
Description: number of ICU days was collected for subjects who received RBX2660 and who were subsequently hospitalized for recurrent CDAD treatment.
Time Frame: 6 months
Population: 31 subjects had evaluable data at 6 months.
Measure: Median (Full Range); unit: number of particpants' ICU days
Arm/Group | RBX2660 (Microbiota Suspension)
Number analyzed (Participants) | 31
number of particpants' ICU days | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: From time of enrollment through the 6-month follow-up period.
Arm/Group | RBX2660 (Microbiota Suspension)
Serious Adverse Events (participants affected / at risk) | 7/34
Other Adverse Events (participants affected / at risk) | 23/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBX2660 (Microbiota Suspension) (N=34)
Clostridium difficile infection (Infections and infestations) | 3 (4)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Clostridium difficile Colitis (Infections and infestations) | 1 (3)
Bacteraemia (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 1 (1)
Chemotherapy (Surgical and medical procedures) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBX2660 (Microbiota Suspension) (N=34)
Abdominal Distension (Gastrointestinal disorders) | 7 (9) — Most were mild-moderate in severity and resolved within 7 days of receiving RBX2660.
Abdominal Pain (Gastrointestinal disorders) | 10 (14)
Anorectal Discomfort (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 8 (14)
Diarrhoea (Gastrointestinal disorders) | 10 (26)
Flatulence (Gastrointestinal disorders) | 13 (15)
Nausea (Gastrointestinal disorders) | 5 (5)
Proctalgia (Gastrointestinal disorders) | 2 (3)
Vomiting (Gastrointestinal disorders) | 4 (5)
Chills (General disorders) | 5 (5)
Fatigue (General disorders) | 3 (3)
Pyrexia (General disorders) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (3)
Urinary Tract Infection (Infections and infestations) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Headach (Nervous system disorders) | 2 (3)
Anxiety (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size (n=34) limits extrapolation of results to a larger population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No